CLINICAL TRIAL: NCT00134069
Title: Phase I/II Clinical, Pharmacological, and Biological Study of BAY 43-9006 in Combination With Cetuximab and Irinotecan in Patients With Advanced Colorectal Cancer
Brief Title: Sorafenib, Cetuximab, and Irinotecan in Treating Patients With Advanced or Metastatic Colorectal Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2009-00110; 07-0571 (Other: Colorado Multiple Institutional Review Board); R21CA117125 (NIH); U01CA070095 (NIH)
Record Dates: First submitted 2005-08-22; First posted 2005-08-24 (Estimated); Last update posted 2014-04-16 (Estimated); Status verified 2014-04

CONDITIONS: Recurrent Colon Cancer; Recurrent Rectal Cancer; Stage III Colon Cancer; Stage III Rectal Cancer; Stage IV Colon Cancer; Stage IV Rectal Cancer
MeSH Terms: conditions — Colonic Neoplasms; Rectal Neoplasms | interventions — Sorafenib; Cetuximab; Irinotecan

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Treatment (sorafenib, irinotecan, cetuximab) (Experimental): Patients will receive sorafenib by mouth once or twice a day and a 1- to 2-hour infusion of cetuximab once a week for 8 weeks. They will also receive a 1½-hour infusion of irinotecan once a week in weeks 3-6. Patients will then receive sorafenib by mouth once or twice a day and a 1- to 2-hour infusion of cetuximab once a week for 6 weeks. They will also receive a 1½-hour infusion of irinotecan once a week in weeks 1-4. Treatment may repeat every 6 weeks for as long as benefit is shown.
  Interventions: Drug: sorafenib tosylate; Drug: cetuximab; Drug: irinotecan hydrochloride

INTERVENTIONS:
Drug: sorafenib tosylate — Given orally
  Other Names: BAY 43-9006; BAY 43-9006 Tosylate Salt; BAY 54-9085; Nexavar; SFN
Drug: cetuximab — Given IV
  Other Names: C225; C225 monoclonal antibody; IMC-C225; MOAB C225; monoclonal antibody C225
Drug: irinotecan hydrochloride — Given IV
  Other Names: Campto; Camptosar; CPT-11; irinotecan; U-101440E

SUMMARY:
This phase I/II trial is studying the side effects and best dose of sorafenib when given together with cetuximab and irinotecan and to see how well they work in treating patients with advanced or metastatic colorectal cancer. Sorafenib may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth. Monoclonal antibodies, such as cetuximab, can block tumor growth in different ways. Some block the ability of tumor cells to grow and spread. Others find tumor cells and help kill them or carry tumor-killing substances to them. Sorafenib and cetuximab may also stop tumor growth by blocking blood flow to the tumor. Drugs used in chemotherapy, such as irinotecan, work in different ways to kill tumor cells, either by killing the cells or by stopping them from dividing. Giving sorafenib together with cetuximab and irinotecan may kill more tumor cells

DETAILED DESCRIPTION:
OBJECTIVES:

I. Determine the toxicity spectrum and dose-limiting toxic effects of sorafenib when combined with cetuximab and irinotecan in patients with advanced or metastatic colorectal cancer.

II. Determine the recommended phase II dose of sorafenib when combined with cetuximab and irinotecan in these patients.

III. Correlate the clinical activity of this regimen, in terms of radiologic and positron emission tomography (PET) response, with baseline extracellular signal-regulated kinase (ERK) expression as well as Kirsten rat sarcoma (KRAS), BRAF, and other genetic properties of tumors in these patients.

IV. Determine the pharmacokinetics of this regimen in these patients. V. Correlate the pharmacodynamic effects of this regimen with baseline ERK expression as well as KRAS, BRAF, and other genetic properties of tumors in these patients.

VI. Correlate the pharmacodynamic effects of this regimen on mitogen-activated protein kinase (MAPK) status in peripheral blood mononuclear cells and on normal skin and oral mucosa with clinical parameters in these patients.

OUTLINE: This is a phase I dose-escalation study of sorafenib followed by a multicenter phase II study.

PHASE I:

COURSE 1 (56 days): Patients receive oral sorafenib once or twice daily on days 1-56, cetuximab IV over 1-2 hours on days 1, 8,15, 22, 29, 36, 43, and 50, and irinotecan IV over 90 minutes on days 15, 22, 29, and 36.

COURSE 2 AND ALL SUBSEQUENT COURSES (42 days): Patients receive oral sorafenib once or twice daily on days 1-42, cetuximab IV over 1-2 hours on days 1, 8, 15, 22, 29, and 36, and irinotecan IV over 90 minutes on days 1, 8, 15, and 22. Courses repeat every 42 days in the absence of disease progression or unacceptable toxicity.

Cohorts of 3-6 patients receive escalating doses of sorafenib until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose preceding that at which 2 of 3 or 2 of 6 patients experience dose-limiting toxicity. At least 6 patients are treated at the MTD.

PHASE II: Patients receive sorafenib at the MTD determined in phase I, cetuximab, and irinotecan as in phase I.

After completion of study treatment, patients are followed at 30 days.

*NOTE: This trial was intended to be Phase I/II, but the trial never continued to the Phase II portion.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed colorectal cancer (advanced or metastatic disease not amenable to potential curative resection)
* Archival tumor (blocks and/or slides) must be available for patients who decline tumor biopsies
* Tumor must be amenable to sequential biopsies for patients willing to undergo tumor biopsy
* Must have evidence of disease progression after first-line chemotherapy for advanced disease
* Previously irradiated lesions are not considered measurable disease
* Measurable disease, defined as >= 1 unidimensionally measurable target lesion >= 20 mm by conventional techniques OR >= 10 mm by spiral CT scan
* No known brain metastases
* Eastern Cooperative Oncology Group (ECOG) 0-2 OR Karnofsky 60-100%
* Life expectancy of more than 12 weeks
* white blood cell count (WBC) >= 3,000/mm^3
* Bilirubin normal
* Creatinine normal OR creatinine clearance >= 60 mL/min
* No hypertension
* No symptomatic congestive heart failure
* No unstable angina pectoris
* No cardiac arrhythmia
* Not pregnant or nursing
* Able to swallow oral medication
* Willing to undergo 2 sequential tumor and skin biopsies
* No ongoing or active infection
* No history of allergic reaction attributed to compounds of similar chemical or biologic composition to study drugs
* No psychiatric illness or social situation that would preclude study compliance
* No other uncontrolled illness
* No prior cetuximab
* No concurrent prophylactic filgrastim (G-CSF), sargramostim (GM-CSF) or epoetin alfa
* At least 4 weeks since prior chemotherapy (6 weeks for nitrosoureas or mitomycin) and recovered
* No other concurrent chemotherapy
* More than 4 weeks since prior radiotherapy and recovered
* No prior sorafenib
* No other prior therapy targeted against MAPK
* More than 14 days since prior and no concurrent administration of the following cytochrome P450 3A4 (CYP3A4) inducers:

  * Rifampin
  * Rifabutin
  * Hypericum perforatum (St. John's wort)
  * Phenytoin
  * Carbamazepine
  * Phenobarbital
* More than 7 days since prior and no concurrent administration of the following CYP3A4 inhibitors:

  * Amiodarone
  * Clarithromycin
  * Diltiazem
  * Erythromycin
  * Grapefruit juice
  * Indinavir
  * Saquinavir
  * Lopinavir in combination with ritonavir
  * Fosamprenavir
  * Ritonavir
  * Atazanavir
  * Nelfinavir
  * Itraconazole
  * Ketoconazole
  * Nefazodone
* No concurrent combination antiretroviral therapy for HIV-positive patients
* No other concurrent investigational agents
* No other concurrent anticancer therapy
* Negative pregnancy test
* Fertile patients must use effective contraception
* Absolute neutrophil count >=1,500/mm^3
* Platelet count ≥ 100,000/mm^3
* No evidence of bleeding diathesis
* Aspartate aminotransferase (AST) and Alanine Aminotransferase (ALT) ≤ 2.5 times upper limit of normal

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2005-06; Primary Completion 2010-09 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
Toxicity spectrum and dose-limiting toxicities of sorafenib in combination with cetuximab and irinotecan as assessed by NCI Common Toxicity Criteria for Adverse Effects (CTCAE) v 3.0 | Up to 30 days
Recommended dose for phase II evaluation of the combination of sorafenib, cetuximab and irinotecan | 56 days
Clinical activity of the combination of sorafenib, cetuximab and irinotecan in terms of radiological response | Up to 30 days
Pharmacokinetics of sorafenib, cetuximab, and irinotecan when given in combination or when given in combination with cetuximab alone and with cetuximab and irinotecan | Up to 30 days
Pharmacodynamics of the combination of irinotecan when given in combination with sorafenib and cetuximab in tumor tissues | Up to 30 days

CONTACTS AND LOCATIONS:
Overall Officials: Wells Messersmith, Principal Investigator — University of Colorado at Denver Health Sciences Center
Locations (2):
- United States (2):
  - University of Colorado at Denver Health Sciences Center, Aurora, Colorado
  - Johns Hopkins University, Baltimore, Maryland